CLINICAL TRIAL: NCT01274377
Title: A Pilot Trial of CMV Specific Donor Lymphocyte Infusions From 3-6/6 HLA Matched Family Member Following Nonmyeloablative Allogeneic Stem Cell Transplantation
Brief Title: Trial of CMV Specific DLIs From 3-6/6 HLA Matched Family Member Following Nonmyeloablative Allo SCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Nelson Chao (Other)
Responsible Party: Sponsor-Investigator, Nelson Chao, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00013947
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Cytomegalovirus Infections
Keywords: nonmyeloablative allogeneic stem cell transplantation; cytomegalovirus; donor lymphocyte infusions; cytotoxic T lymphocyte
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recipients Using 3-5/6 Matched Donors (Experimental): There will be an equal number of subjects (10) receiving transplants from 3-5/6 Human Leukocyte Antigen (HLA) Matched Donors as those receiving transplants from 6/6 HLA Matched Donors for a total of 20 subjects on study.
  Interventions: Biological: CMV Specific T Cell donor lymphocyte infusion
- Recipients Using 6/6 Matched Donors (Experimental): There will be an equal number of subjects (10) receiving transplants from 3-5/6 HLA Matched Donors as those receiving transplants from 6/6 HLA Matched Donors for a total of 20 subjects on study.
  Interventions: Biological: CMV Specific T Cell donor lymphocyte infusion

INTERVENTIONS:
Biological: CMV Specific T Cell donor lymphocyte infusion — Donor Lymphocyte Infusion (DLI)
  Other Names: Miltenyi Biotec

SUMMARY:
Human cytomegalovirus (CMV) is a benign infectious agent in the normal host, but in immunocompromised individuals, such as recipients of stem cell transplants, this virus is a major cause of morbidity and mortality. While pharmacologic agents exist to treat CMV disease, these medications have numerous side effects, the most serious of which is myelosuppression. The frequency of neutropenia ranges from 41% to 58% in stem cell transplant (SCT) patients treated with ganciclovir. Withdrawal of anti-CMV therapy due to these complications may result in recurrent disease. The restoration of cellular immunity to CMV is necessary in order to prevent viral reactivation, and the generation of cytotoxic T cells against CMV early antigens is perhaps the most important part of the host immune response to CMV. At day 40 post-transplant, for example, at least 65% of SCT patients are deficient in CD8+ T-cell responses to CMV. Previous studies have demonstrated a direct correlation between CMV infection in these patients and cytotoxic T lymphocyte (CTL) function, with patients who have defects in cellular immunity being at high risk for invasive CMV disease. The median time post-transplant for the development of CMV disease is 50 to 60 days, and CMV re-activation occurs in 70 to 80% of CMV sero-positive SCT recipients. Without anti-viral therapy as many as 50% of these patients will develop CMV disease.

DETAILED DESCRIPTION:
This protocol will evaluate the safety of CMV specific T cell infusion following nonmyeloablative stem cell transplantation from 3-6/6 HLA matched donors as well as evaluate the efficacy of antigen specific T cell infusions in preventing CMV activation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have undergone a non-myeloablative allogeneic transplant, using a 3-6/6 Human Leukocyte Antigen (HLA) matched related donor.
2. Subjects must be CMV seropositive prior to transplant by CMV immune screen or CMV IgG or develop detectable disease by PCR in the post-transplant setting.
3. Performance status must be Karnofsky 50-100%.
4. Donor cellular engraftment of at least 2.5% from the non-myeloablative procedure and prior to the first infusion.
5. ≤ Grade 1 acute graft versus host disease (GVHD) at time of the CMV specific T cell infusion. Patients with treated acute GVHD must be on a stable dose of therapy (no increase in immunosuppressive therapy for the 2 weeks before planned donor cell infusion). The dosage level of immunosuppressive therapy at the time of infusion should be no greater than 20 mg of prednisone daily or mycophenolate 1000 mg tid daily or cyclosporine with a target level of 200 ng/ml or equivalent.
6. At the time of the CMV specific T cell infusion, the recipient must have adequate organ function as indicated by < Grade 3 across all organ systems except for hematologic toxicity.
7. Subject must be at least 18 years of age.

Exclusion Criteria:

1. Pregnant or lactating women,
2. Subjects with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise compliance with this protocol.
3. Subjects who had histopathologically confirmed overall Grade 4 GVHD lasting longer than 7 days, from the non-myeloablative therapy, are not eligible.

Donor Inclusion/Exclusion Criteria

1. Adult donors must be the same donor used for the non-myeloablative allogeneic transplant and must be a related family member with a HLA 3-6/6 match with the subject and must be capable of providing informed consent; Potential donors under the age of 18 must have a 'single patient exemption' approved by the Institutional Review Board (IRB) and the donor and a guardian must provide assent. The donor must be the same donor used for the original allogeneic transplantation. Selection of donors will be compliant with 21 CFR 1271.
2. Adult donors must be CMV seropositive prior to transplant by CMV immune screen or CMV IgG positive.
3. Donors will complete the Adult Donor History Questionnaire and have all laboratory studies included in the Donor Referral NTL Panel, CBC with auto or manual differential, and a Chemistry Panel within 7 days of scheduled collection procedure. Donors who were evaluated greater than 1 year prior for transplant collection will also have a history and Physical Exam, CXR, and EKG completed. Donors must not have any medical condition which would make apheresis more than a minimal risk, and should have normal range laboratory findings. All abnormal laboratory findings will be evaluated by the treating physician within the context of the entire donor assessment process.
4. Females of childbearing potential should have a negative serum beta-HCG (human chorionic gonadotropin) test within 1 week of beginning apheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02-23 (Actual); Study Completion 2015-10-05 (Actual)

PRIMARY OUTCOMES:
Safety of CMV Specific T cell infusion following Stem Cell Transplant | 2 years
  Donor Lymphocyte Infusion (DLI) of CMV Specific T cell clones following nonmyeloablative allogeneic stem cell transplant for the prevention of CMV

SECONDARY OUTCOMES:
Efficacy of CMV-specific T cell infusion in terms of response, progression free survival, and overall survival | 2 years
  The efficacy and its effect on survivability will be assessed.
Evaluate the recovery of immune function post engraftment with this regimen. | 2 years
  Blood samples will be collected for immune reconstitution studies, including assessing CMV specific responses, just prior to each cell infusion, and 3,6, 12 months post last infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Chao, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States